CLINICAL TRIAL: NCT06897345
Title: Comparison of Postoperative Analgesic Efficacy of Transversus Abdominis Plan Block and Rectus Sheath Block in Abdominoplasty Cases: A Randomized Prospective Clinical Trial
Brief Title: Transversus Abdominis Plan Block Versus Rectus Sheath Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aysel Salkaya, Anesthesiologist, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: salkaya-1
Record Dates: First submitted 2025-03-13; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Abdominal Obesity; Postoperative Pain; Postoperative Complications
Keywords: post operative pain; transversus abdominis plane block; rectus sheat block
MeSH Terms: conditions — Obesity, Abdominal; Pain, Postoperative; Postoperative Complications

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transversus abdominis plane block (Active Comparator): After administering 0.02 mg/kg midazolam for sedation to Group TAP patients, they will be placed in the supine position on both sides under sterile conditions using the high-frequency linear probe of the Esaote CA631 brand ultrasound, and the linear probe will be slid from the bilateral umblicus level to the midaxillary line, and when the internal and external oblique muscles are seen, the needle will be advanced from medial to lateral in an inplane manner, and the fascia between the internal oblique and transversus abdominis muscles will be reached, and after negative aspiration, 20 cc of 0.25% bubivacaine will be injected.
  Interventions: Procedure: transversus abdominis plane block
- rectus sheat block (Active Comparator): After administering 0.02 mg/kg midazolam for sedation, in the supine position, under sterile conditions, using the high-frequency linear probe of the Esaote CA631 brand ultrasound, 1 cm laterally over the umblicus, and after negative aspiration between the rectus muscle and the posterior rectus sheath, 20 cc of 0.25% bubivacaine will be injected (bilateral). 15 minutes after the block is applied, general anesthesia will be applied to the patients in both groups with 1 mcg/kg fentanyl, 2 mg/kg propofol, 0.6 mg/kg rocuronium intravenously and they will be orotracheal intubated. Intraoperative remifentanil needs will be recorded. Within the scope of multimodal analgesia, 1 g paracetamol will be administered to all patients 30 minutes before the end of the operation and 3 mg/kg sugammadex will be administered at the end of the operation and they will be extubated.
  Interventions: Procedure: rectus sheat block

INTERVENTIONS:
Procedure: transversus abdominis plane block — The transversus abdominis plane (TAP) block is a regional anesthesia technique used primarily to provide pain relief for patients undergoing surgery in the abdominal region. The TAP block targets the nerves that supply sensations to the skin and muscles of the abdominal wall.
  Other Names: bupivakain
  Arms: transversus abdominis plane block
Procedure: rectus sheat block — The rectus sheath block is a type of regional anesthesia used primarily for pain management in the abdominal area. It involves injecting local anesthetic into the rectus sheath, which is the fibrous sheath that envelops the rectus abdominis muscle. This block targets the lower intercostal nerves as they traverse through the sheath, thereby providing analgesia to the anterior abdominal wall.
  Other Names: bupivakain
  Arms: rectus sheat block

SUMMARY:
The investigator aims to compare the analgesic efficacy of Transversus Abdominis Plan Block and Rectus Sheath Block which are used to prevent intraoperative and postoperative pain and reduce the use of opioid in abdominoplasty operations.

DETAILED DESCRIPTION:
Abdominoplasty is a frequently performed surgical procedure in aesthetic and plastic surgery. It is performed to solve the pain caused by the large abdomen, respiratory distress and aesthetic problems. Since large tissue excision is made and a large area is worked on, providing perioperative pain control is also important to prevent both postoperative respiratory distress and postoperative chronic pain formation.

In order to prevent both intraoperative and postoperative pain and to reduce opioid use, peripheral nerve blocks that provide analgesia on the abdominal wall can be applied to patients before the surgical incision. The most well-known of these blocks is the Transversus Abdominis Plane block. Another block that has been proven effective in abdominal surgery is the Rectus Sheath block. In the Transversus Abdominis Plane block (TAP), local anesthetic is injected into the fascia between the internal oblique and transversus abdominis muscles, aiming for analgesia. It provides multidermatomal sensory block by spreading the local anesthetic agent in the fascial area. The Rectus Sheath (RK) block is also a preferred plan block in abdominoplasty surgery. In this block, local anesthetic agent is injected between the rectus muscle and the posterior rectus sheath to achieve analgesia.

Although the effectiveness of both blocks has been shown mostly in abdominoplasty operations, there is no publication in the literature showing and comparing their effectiveness in abdominoplasty operations. With this study, The investigator aimed to compare the analgesic effectiveness of the two blocks in patients who will undergo abdominoplasty operations.

ELIGIBILITY:
Inclusion Criteria:

Patients who will undergo elective abdominoplasty

* Patients between the ages of 18-65
* ASA (American Society of Anesthesiologists) I-II-III patients
* Patients with a body weight between 50-80 kg

Exclusion Criteria:

* - ASA IV patient group
* Patients under 18 years of age
* Patients without cooperation
* Patients with chronic alcohol use
* Patients in whom peripheral plane block application is contraindicated (infection at the application site, coagulopathy, local anesthetic allergy)
* Patients who do not want to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | VAS scores were measured at the beginning, st, 3rd, 6th, 12th and 24th hour in the postoperative recovery unit.
  The Visual Analog Scale (VAS) score is a subjective measurement tool used to assess the intensity of pain. It is commonly used in clinical settings to help patients communicate their pain levels to healthcare providers. The VAS typically consists of a straight line, often 10 centimeters long, with one end labeled "no pain" (0) and the other end labeled "worst pain imaginable" (10). Patients mark a point on the line that corresponds to their current level of pain.

SECONDARY OUTCOMES:
total analgesic consumption | 24 hour
  Total analgesic consumption of patients in the first 24 hours postoperatively
first analgesic need | 24 hour
  Time until first postoperative analgesic requirement

CONTACTS AND LOCATIONS:
Overall Officials: LEYLA KILINC, Study Chair — şişli etfal eğitim araştırma hastanesi
Locations (1):
- Sisli Hamidiye Etfal Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No